CLINICAL TRIAL: NCT03977363
Title: The Portuguese Survey on Anticoagulated Patients Register (START-Portugal-Register)
Acronym: START-Portugal
Status: Terminated | Type: Observational
Why Stopped: Halted Prematurely
Sponsor: CHAD (Other)
Responsible Party: Sponsor-Investigator, CHAD, Prof. Francisco Batel Marques, Association for Innovation and Biomedical Research on Light and Image
Organization: Association for Innovation and Biomedical Research on Light and Image (Other)
Other Study IDs: CHAD-2019-01
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Heart Valve Diseases or Prosthesis
Keywords: Anticoagulation; Anticoagulants; Vitamin K antagonists; Warfarin; Low molecular weight heparin; Direct oral anticoagulants; dabigatran; rivaroxaban; apixaban; edoxaban; Atrial Fibrillation; Thromboembolism; Venous Thromboembolism; Heart Valve Diseases; Arrhythmia; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Embolism and Thrombosis
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism; Heart Valve Diseases; Thromboembolism; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Vascular Diseases; Embolism and Thrombosis | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Anticoagulated patients: Patients receiving anticoagulation treatment
  Interventions: Drug: Anticoagulant drugs

INTERVENTIONS:
Drug: Anticoagulant drugs — Anticoagulant drugs

SUMMARY:
Anticoagulants are used to prevent thrombotic events in patients with predisposing factors. However, the use of such therapies is associated with bleeding complications, which can be a serious safety issue. Thus, it is important to evaluate the safety and effectiveness of such therapies based on data collected in clinical practice in order to generate relevant scientific data that could be used to support clinical and regulatory decisions.

This is an open, prospective, multicenter, observational cohort study that aims to prospectively record the clinical history of adult patients receiving anticoagulant treatment, irrespectively of the prescribed drug and the indication for its use.

DETAILED DESCRIPTION:
* The Portuguese Survey on anTicoagulated pAtients RegisTer (START-Portugal-Register) is an open, prospective, multicenter, observational cohort study that intends to record the clinical history of adult patients receiving anticoagulant therapies, providing real-world data on the safety and effectiveness of such therapies, as well as to serve as the starting point of collaborative clinical studies, enabling their planning and execution.
* The START-Portugal-Register is designed solely for observational purposes; it is not intended to have any influence on the treatment of included patients.
* Objectives:

  * To prospectively record the clinical history of adult patients receiving anticoagulant treatment, irrespectively of the prescribed drug and the indication for its use.
  * To enhance the understanding of risks and benefits associated with the use of anticoagulant drugs in routine clinical practice;
  * To prospectively record decisions and reasons guiding physicians' decisions in order to manage anticoagulant treatment options in routine clinical practice;
  * To improve knowledge on the epidemiologic, diagnostic and clinical features of thrombotic diseases;
  * To generate real-world evidence on the safety and effectiveness of anticoagulant drugs, therefore contributing to support informed clinical decisions.
* The START-Portugal-Register is open to the participation of clinical centers and individual physicians that are involved in the management of patients undergoing anticoagulant treatment.
* Patients who sign the informed consent and fulfil the inclusion/exclusion criteria will be enrolled in the study and considered for data analysis.
* Follow-up: mandatory for at least 12 months. Nevertheless, a long-term follow-up is recommended for patients who receive an indefinite anticoagulation treatment. The START-Portugal-Register sets itself an indefinite time limit.
* A descriptive analysis will be conducted for all study variables. A propensity score model will be applied to compare the safety and efficacy of the different anticoagulant treatments.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Patients who, at the time of inclusion, have been receiving for no more than 30 days or are about to start anticoagulation therapy - irrespectively of the prescribed drug, the dosage, and the indication for its use;
* Availability to sign an informed consent form.

Exclusion Criteria:

* Not available for follow-up and constant monitoring;
* Participation in phase II or III clinical studies*;
* Life-expectancy <6 months, non-residents in the Participant region, or planning to leave in the next 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The START-Portugal-Register is open to the participation of clinical centers and individual physicians (called Participants) that are involved in the management of patients undergoing anticoagulant treatment. Participants are required to enroll patients consecutively, without any a-priori exclusion criteria other than life-expectancy,lack of availability for follow-up or geographical inaccessibility.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Incidence of complications | At least 12 months of follow-up
  From date of inclusion in the registry until the date of first documented complication or date of death from any cause, whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Batel Marques, PhD, Principal Investigator — AIBILI - Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI - Association for Innovation and Biomedical Research on Light and Image, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Testa S, Paoletti O, Zimmermann A, Bassi L, Zambelli S, Cancellieri E. The role of anticoagulation clinics in the era of new oral anticoagulants. Thrombosis. 2012;2012:835356. doi: 10.1155/2012/835356. Epub 2012 Oct 14. PMID 23097696
- [Background] Antonucci E, Poli D, Tosetto A, Pengo V, Tripodi A, Magrini N, Marongiu F, Palareti G; START-Register. The Italian START-Register on Anticoagulation with Focus on Atrial Fibrillation. PLoS One. 2015 May 22;10(5):e0124719. doi: 10.1371/journal.pone.0124719. eCollection 2015. PMID 26001109
- [Background] Ruff CT, Giugliano RP, Braunwald E, Hoffman EB, Deenadayalu N, Ezekowitz MD, Camm AJ, Weitz JI, Lewis BS, Parkhomenko A, Yamashita T, Antman EM. Comparison of the efficacy and safety of new oral anticoagulants with warfarin in patients with atrial fibrillation: a meta-analysis of randomised trials. Lancet. 2014 Mar 15;383(9921):955-62. doi: 10.1016/S0140-6736(13)62343-0. Epub 2013 Dec 4. PMID 24315724
- [Background] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Background] Schulman S, Kearon C, Kakkar AK, Mismetti P, Schellong S, Eriksson H, Baanstra D, Schnee J, Goldhaber SZ; RE-COVER Study Group. Dabigatran versus warfarin in the treatment of acute venous thromboembolism. N Engl J Med. 2009 Dec 10;361(24):2342-52. doi: 10.1056/NEJMoa0906598. PMID 19966341
- [Background] Agnelli G, Buller HR, Cohen A, Curto M, Gallus AS, Johnson M, Porcari A, Raskob GE, Weitz JI; AMPLIFY-EXT Investigators. Apixaban for extended treatment of venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):699-708. doi: 10.1056/NEJMoa1207541. Epub 2012 Dec 8. PMID 23216615
- [Background] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658
- [Background] Caldeira D, Rodrigues FB, Barra M, Santos AT, de Abreu D, Goncalves N, Pinto FJ, Ferreira JJ, Costa J. Non-vitamin K antagonist oral anticoagulants and major bleeding-related fatality in patients with atrial fibrillation and venous thromboembolism: a systematic review and meta-analysis. Heart. 2015 Aug;101(15):1204-11. doi: 10.1136/heartjnl-2015-307489. Epub 2015 Jun 2. PMID 26037103
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354